CLINICAL TRIAL: NCT04691739
Title: Teletherapy for Upper Extremity Fracture Rehabilitation, A Pilot Randomized Controlled Trial (TELE-REHAB Study)
Brief Title: Teletherapy for Upper Extremity Fracture Rehabilitation (TELE-REHAB Study)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not enroll participants that meet inclusion criteria outlined in the study protocol. All screening and enrollment attempts have ended.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Christopher Langhammer, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00094373
Record Dates: First submitted 2020-12-24; First posted 2020-12-31 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Upper Limb Surgery; Occupational Therapy
Keywords: Upper Limb Surgery; Upper Extremity Injury; Occupational Therapy
MeSH Terms: conditions — Arm Injuries | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person occupational therapy (Active Comparator): occupational therapy delivered in-person
  Interventions: Other: occupational therapy
- Teletherapy (Active Comparator): Video-conferencing occupational therapy
  Interventions: Other: occupational therapy

INTERVENTIONS:
Other: occupational therapy — occupational therapy sessions include a set of standardized test exercises plus additional modalities that are optimized to each patient's needs according to the clinical judgement of the treating therapist

SUMMARY:
Following upper limb surgeries, patients could receive occupational therapy either in-person or remotely (teletherapy). The investigators currently do not know which occupational therapy delivery is better in terms of clinical outcomes and patient recovery. The proposed study is a pilot randomized controlled trial (RCT) testing the feasibility of comparing in-person occupational therapy to teletherapy following operative fixation of upper extremity fracture. It is a single site, parallel-arm, randomized controlled trial to compare teletherapy versus in-person occupational therapy. Patients who are eligible will be randomized similar to a flip of a coin (1:1) to occupational therapy in-person or through a telemedicine platform. Patients would also complete surveys at each follow-up visit to measure clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had operative fixation of upper extremity fracture located between the humeral shaft and distal radius (inclusive) who are indicated for outpatient occupational therapy.
* Participants at least 18 years (≥ 18 years of age).
* English-speaking participants

Exclusion Criteria:

* Participants unable to consent
* Vulnerable populations including prisoners and marginally housed patients
* Additional traumatic conditions that may affect the ultimate-use pattern of the injured limb including traumatic brain injury, spinal cord injury, peripheral nerve injury, or associated soft tissue injury requiring specific postoperative activity modifications.
* Contralateral upper extremity injury that prevents participating in the standardized exercises.
* Initiation of occupational therapy (OT) during an inpatient hospital stay
* Pre-existing comorbidities that may interfere with communication or that may limit the use of standard telecommunications tools (sight/hearing impaired, speech impaired)
* Patients without a smart-phone or internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome 1: Enrollment rate | At 12 months
  A success threshold of 40% enrollment of eligible patients
Feasibility outcome 2a: Completion rate | at 6 weeks
  A success threshold of 90% patient follow-up and case report forms completion rates
Feasibility outcome 2b: Completion rate | at 3 months
  A success threshold of 90% patient follow-up and case report forms
Feasibility outcome 2c: Completion rate | at 6 months
  A success threshold of 90% patient follow-up and case report forms

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Langhammer, MD, Principal Investigator — U of Maryland, Baltimore
Locations (1):
- U of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No